CLINICAL TRIAL: NCT07205588
Title: RESTODATA-NUM: A Multicenter Observational Study on the Assessment of Dental Pathologies Using Digital Tools in Adults
Brief Title: Assessment of Dental Pathologies Using Digital Tools
Acronym: RESTODATA-NUM
Status: Recruiting | Type: Observational
Sponsor: Recherche Clinique en Odontologie (ReCOL) (Network)
Responsible Party: Sponsor
Other Study IDs: RECOL 2024-01
Record Dates: First submitted 2025-07-17; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries (Diagnosis); Dental Plaque (Diagnosis); Periodontitis
MeSH Terms: conditions — Dental Caries; Disease; Dental Plaque; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Digital technology is playing an increasingly important role in dentistry, because of its ability to support the practitioner and increase work efficiency.

Among digital tools, orthopantomogram (OPT or panoramic) radiography is currently the most widely used. It provides a global view of the jaws, highlighting internal structures in 2D.

As in other fields, scientific advances have made it possible to go beyond the limited representation of two planes of space and obtain 3D images.

The intraoral scanner (IOS) or "optical impression camera" appeared in the mid-80s. They use light to create a digital optical impression that reproduces the surface of external anatomical structures in 3D images. It improves dental practice, making impressions less uncomfortable for patients, saving clinical time, facilitating storage and archiving, and facilitating transmission to the prosthetist where appropriate. This type of device is already well established in dental practices.

More recently, Cone Beam Computed Tomography (CBCT) has also begun to develop. This 3D sectional imaging technique adds an extra dimension to the exploration of internal structures.

Imaging examinations provide additional information to that obtained from the visual clinical oral examination. Together, they help the practitioner to establish the diagnosis and treatment plan.

Currently, visual information has to be collected manually. Collecting this data represents a significant amount of information. Its quality and completeness are crucial to the success of the treatment.

Given the high volume of consultations, and practitioners' need to optimize their time, it would be interesting to assess whether optical impressions, at least in part, could help to acquire this clinical data more systematically and more rapidly, in order to improve patient management.

Similarly, Cone Beam CT (CBCT), with its 3D data, improves the accuracy of diagnostic information. It would also be interesting to assess the real added value of this examination.

The RESTODATA-NUM study follows on from the RESTODATA study, the results of which provided recent information on the oral status of adult patients, and their care needs.

The aim of this study is to compare the performance of a standard real-life examination by the practitioner combining clinical and radiographic examinations (referred to here as practitioner-on-patient detection) on the one hand, and an examination based on imaging results obtained using digital tools on the other, in terms of detecting dental condition in a sample of adult patients consulting for an oral examination at one of the participating centers.

DETAILED DESCRIPTION:
Digital technology is playing an increasingly important role in dentistry due to its ability to assist practitioners and enhance work efficiency.

Among digital tools, panoramic radiography (orthopantomogram) is currently the most widely used. It provides a comprehensive image of the jaws, highlighting internal structures in 2D. As in other fields, scientific advances have made it possible to go beyond two-dimensional representations and obtain 3D images.

The intraoral scanner, also known as an "optical impression camera," emerged in the mid-1980s. These devices use light to create a digital optical impression that reproduces the surface of external anatomical structures in 3D images. They improve dental practice by making impression-taking less uncomfortable for patients, saving clinical time, simplifying storage and archiving, and facilitating transmission to dental technicians when needed. This type of device is already well established in dental practices.

More recently, Cone Beam Computed Tomography (CBCT), also known as digital volumetric tomography with a conical beam, has begun to develop. This 3D sectional imaging technique allows for the exploration of internal structures by adding an extra dimension.

Imaging examinations provide additional information that complements the findings of the visual clinical oral examination. Together, they help the practitioner establish a diagnosis and treatment plan. Currently, visual information must be recorded manually. Collecting this data represents a significant amount of information, and the success of treatment partly depends on its quality and completeness.

Given the high volume of consultations and the need for practitioners to optimize their time, it would be worthwhile to assess whether optical impressions could help systematically and quickly acquire some of this clinical data to improve patient care.

Similarly, the 3D data provided by CBCT enhances the accuracy of diagnostic information. It would also be useful to evaluate the actual added value of this examination.

The RESTODATA-NUM study follows on from the RESTODATA study, whose results provided recent insights into the oral health status and care needs of adult patients.

The objective of this study is to compare the performance of a standard real-life examination by a practitioner-combining clinical and radiographic assessments-with an examination based on imaging results obtained using digital tools, in terms of detecting dental conditions in a sample of adult patients undergoing an oral examination at one of the participating centers.

Information on the Type of Clinical Investigation:

This is an observational, descriptive, and multicenter study. Based on these characteristics, the study is initially classified by the principal investigator as a Category 3 research project under the Jardé Law (Article R1121-3 of the French Public Health Code, Decree No. 2006-477 of April 26, 2006). The digital tools used in this study (intraoral scanner, panoramic radiography, and cone beam computed tomography) are routinely employed in dental practices. Radiographs will only be performed when medically justified. There will be no deviation from standard patient care, and no additional procedures will be introduced.

Overview of the ReCOL Network and Participating Private Practices:

The ReCOL network is a French clinical research network in dentistry, inspired by a similar model in the United States. Its goal is to involve private dental practitioners in clinical studies. Established in 2018, ReCOL has already conducted several studies, many of which are available on its website: https://recol.fr. The network operates collaboratively, with research topics discussed within the association's executive board. The idea for the RESTODATA-NUM study emerged from one of these discussions.

A total of 36 dental surgeons, all equipped with the necessary tools for the study, responded positively to a call for participation sent via email to all ReCOL members. Some of these practitioners had previously participated in the RESTODATA study.

Study Procedure and Data Collection:

Each participant will attend a single study visit.

Eligibility will be assessed by the investigating dental surgeon. The study will be offered to all patients attending a participating center for an oral examination who meet the inclusion criteria.

An information letter will be provided to each patient. If no urgent care is required, patients may take up to seven days to consider participation and reschedule their appointment if desired. Upon agreement, the patient will sign a non-opposition form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have read the information sheet and agreed to participate in the study
* Patients affiliated with a social security scheme
* Patients aged 18 years or older
* New patients to the practice or patients who have not visited the practice in the past six months

Exclusion Criteria:

* Patient who has expressed opposition to participating in the study
* Age < 18 years
* Individual under legal guardianship or curatorship
* Pregnant woman
* Patient currently undergoing orthodontic treatment with fixed appliances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to all patients attending a participating investigation center for an oral examination who meet the study's inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Decayed, Missing, or Filled Teeth in the permanent dentition, measured both clinically and from intraoral scan (IOS) images using the DMFT index | at the day of the dental examination
  Number of Decayed, Missing, or Filled Teeth in the permanent dentition, measured both clinically and from intraoral scan (IOS) images using the DMFT index

SECONDARY OUTCOMES:
Location and extent of carious dental lesions | At the day of the dental examination
  Location and extent of carious dental lesions:
  Assessed clinically and from intraoral scan (IOS) images using the simplified International Caries Detection and Assessment System, version 6 (ICDAS-6) score, using a scale from 0 to 6. Higher scores indicate worse outcomes, reflecting increasing severity of carious lesions.
  Assessed radiographically on panoramic radiographs (OPT) or cone beam CT (CBCT) using a three-level radiographic scale of carious involvement (enamel, initial dentin, deep dentin)"
Location and extent of dental wear lesions | At the day of the dental examination
  Location and extent of dental wear lesions:
  Assessed clinically and from intraoral scan (IOS) images using the BEWE score Assessed radiographically using a three-level scale of dental tissue thickness reduction (enamel thinning, complete enamel surface loss, enamel surface loss with dentin exposure)
Location, extent, and quality of dental restorations across all detection methods: | At the day of the dental examination
  Location, extent, and quality of dental restorations across all detection methods:
  Assessed based on their type, the number of involved surfaces, and their location (using CCAM coding) Assessed using a three-level index: adequate, minor but acceptable defects (to be monitored), major or harmful defects (requiring repair or replacement)
Periodontal involvement | At the day of the dental examination
  Periodontal involvement (gingival inflammation, presence of calculus, pockets, recession):
  Clinically assessed using the Plaque Index Clinically assessed using the CPITN and DPSI indices Assessed from intraoral scan (IOS) images using a 4-level visual index: healthy, inflammation, inflammation with calculus, inflammation with calculus and recession Radiographically assessed based on the location and severity of bone loss visible on panoramic radiographs (OPT) or cone beam CT (CBCT)
Endodontic status | At the day of the dental examination
  Endodontic status: number and location of teeth with pulpal involvement and periapical complications, detected and assessed radiographically on panoramic radiographs (OPT) or cone beam CT (CBCT):
  Periapical lesion evaluated using the simplified Periapical Index (PAI)
Endodontic status | At the day of the dental examination
  Endodontic status: number and location of teeth with pulpal involvement and periapical complications, detected and assessed radiographically on panoramic radiographs (OPT) or cone beam CT (CBCT):
  Presence of root canal treatment (CCAM code)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Grosgogeat, DDS, PhD, Principal Investigator — Service de Consultations et de Traitements Dentaires Hospices Civils de Lyon
Locations (22):
- France (21):
  - Cabinet dentaire Robbiani, Châtillon
  - AP HP, Colombes
  - Cabinet dentaire Ibn Attya Andaloussi, La Chapelle-sur-Erdre
  - Cabinet dentaire Thiébaut, Landivisiau
  - Cabinet dentaire Lemasson, Latresne
  - Cabinet dentaire Pouchoulin, Les Côtes-d'Arey
  - Cabinet dentaire Dougnac-Galant, Lyon
  - AP HM, Marseille
  - Cabinet dentaire Szerbojm, Ozoir-la-Ferrière
  - Cabinet dentaire Martin, Paimpol
  - Cabinet dentaire Drouhet, Paris
  - Cabinet dentaire Huret, Paris
  - Cabinet dentaire Labidi, Paris
  - Cabinet dentaire Decup, Paris
  - Cabinet dentaire Calvo, Quint-Fonsegrives
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Cabinet cabinet Perier, Saint-Marcellin-en-Forez
  - Cabinet dentaire Guyon-Barras, Saint-Victor-de-Cessieu
  - Cabinet dentaire Delacroix, Thorigné-Fouillard
  - Cabinet dentaire Janisset-Masse, Villiers-sur-Marne
- Cabinet dentaire Enjary, La Saline, Reunion

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Background] Van der Velden U. The Dutch periodontal screening index validation and its application in The Netherlands. J Clin Periodontol. 2009 Dec;36(12):1018-24. doi: 10.1111/j.1600-051X.2009.01495.x. PMID 19929955
- [Background] Ainamo J, Barmes D, Beagrie G, Cutress T, Martin J, Sardo-Infirri J. Development of the World Health Organization (WHO) community periodontal index of treatment needs (CPITN). Int Dent J. 1982 Sep;32(3):281-91. No abstract available. PMID 6958657
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Bartlett D, Ganss C, Lussi A. Basic Erosive Wear Examination (BEWE): a new scoring system for scientific and clinical needs. Clin Oral Investig. 2008 Mar;12 Suppl 1(Suppl 1):S65-8. doi: 10.1007/s00784-007-0181-5. Epub 2008 Jan 29. PMID 18228057
- [Background] Ismail AI, Pitts NB, Tellez M; Authors of International Caries Classification and Management System (ICCMS); Banerjee A, Deery C, Douglas G, Eggertsson H, Ekstrand K, Ellwood R, Gomez J, Jablonski-Momeni A, Kolker J, Longbottom C, Manton D, Martignon S, McGrady M, Rechmann P, Ricketts D, Sohn W, Thompson V, Twetman S, Weyant R, Wolff M, Zandona A. The International Caries Classification and Management System (ICCMS) An Example of a Caries Management Pathway. BMC Oral Health. 2015;15 Suppl 1(Suppl 1):S9. doi: 10.1186/1472-6831-15-S1-S9. Epub 2015 Sep 15. No abstract available. PMID 26391116
- [Background] Decup F, Dantony E, Chevalier C, David A, Garyga V, Tohme M, Gueyffier F, Nony P, Maucort-Boulch D, Grosgogeat B. Needs for re-intervention on restored teeth in adults: a practice-based study. Clin Oral Investig. 2022 Jan;26(1):789-801. doi: 10.1007/s00784-021-04058-5. Epub 2021 Jul 24. PMID 34302555
- [Background] Kaasalainen T, Ekholm M, Siiskonen T, Kortesniemi M. Dental cone beam CT: An updated review. Phys Med. 2021 Aug;88:193-217. doi: 10.1016/j.ejmp.2021.07.007. Epub 2021 Jul 17. PMID 34284332
- [Background] Schmalzl J, Roth I, Borbely J, Hermann P, Vecsei B. The impact of software updates on accuracy of intraoral scanners. BMC Oral Health. 2023 Apr 15;23(1):219. doi: 10.1186/s12903-023-02926-y. PMID 37061664
- [Background] Chi J. Digital Impressions and In-Office CAD/CAM: A Review of Best Practices and What's to Come. Compend Contin Educ Dent. 2021 Mar;42(3):140-141. PMID 34010575